CLINICAL TRIAL: NCT04421001
Title: RCT for Evaluation of Insulin Administration, Time in Range of Glucose, Adverse Events and Quality of Life, While Using the iPORT System in Pediatric Population With Recent-onset Type 1 Diabetes
Brief Title: RCT for Evaluation of Insulin Administration,While Using the iPORT System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0075-20-ASF
Record Dates: First submitted 2020-05-03; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-03

CONDITIONS: T1DM

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- I-Port™*(Medtronic) use Arm (Experimental): Patients will administer insulin via iport system. I-Port™* (Medtronic), infusion set, dedicated for insulin deliery for 72 hours.
  Interventions: Device: I-port use
- Insulin Pen Injections (Active Comparator): Patients will administer insulin via injections as usual
  Interventions: Device: I-port use

INTERVENTIONS:
Device: I-port use — patient will use I-port device fo 2 months

SUMMARY:
Type 1 diabetes is the most common chronic pediatric autoimmune disease, with a rising incidence rate in recent years around the world and in Israel Management includes multiple daily capillary glucose measurements by finger pricks, or interstitial sugar measurements by sensors, and insulin subcutaneous administration before each meal by injections or by an insulin pump .

The initial management and teaching of T1D patients and families includes at least 5-6 glucose measurements per day and at least 4 insulin injections per day, while the preferred guideline should be insulin administration prior to each meal, including morning and afternoon snacks, very common among pediatric patients attending school curriculum.

The early use of I-port at disease diagnosis may reduces pain, increase the amount of daily injections, may increase accuracy of insulin administration, and thus improve time in range from disease diagnosis.

Aims of study:

To assess the efficacy of I-port use in recent onset T1D in a pediatric population, in increasing insulin administration and possibly improving time in range of glucose.

DETAILED DESCRIPTION:
Type 1 diabetes is the most common chronic pediatric autoimmune disease, with a rising incidence rate in recent years around the world and in Israel Management includes multiple daily capillary glucose measurements by finger pricks, or interstitial sugar measurements by sensors, and insulin subcutaneous administration before each meal by injections or by an insulin pump . Treatment goals include several parameters; keeping glucose levels in target range for longer than 70% of the time, having less than 1% of hypoglycemic episodes, and maintaining HbA1c less than 7.5%. In the pediatric population, growth parameters, and quality of life are of major importance in addition. Studies published worldwide in the past decade indicate that only 37% of the diabetic population achieve glycemic control target are balanced with the objective of the glycated hemoglobin (HbA1c) below 7.5%, in all suggested regimens. One of the major obstacles for achieving target goals is the postprandial hyperglycemia. Post prandial hyperglycemia is related to the timing of insulin administration and to the amount injected according to carbohydrate content of the meal A significant association has been demonstrated between missed insulin boluses prior to meals and glycemic control parameters The initial management and teaching of T1D patients and families includes at least 5-6 glucose measurements per day and at least 4 insulin injections per day, while the preferred guideline should be insulin administration prior to each meal, including morning and afternoon snacks, very common among pediatric patients attending school curriculum. The reason for those recommendations is based on quality of life consideration, increasing adherence to management by less daily painful injections. According to ISPAD recommendations, when using injections, it is suggested to consider the use of a device as Insuflon (Unomedical) or I-Port (Medtronic) in order to decrease pain, and enable flexibility of boluses13.

The I-Port system (Medtronic) is intended to allow insulin delivery through the port for 72 hours after port insertion, with one injection, without additional injections or pain. Any insulin, including several types of insulin is delivered via the same port by using the standard insulin pens. The use of I-port system may solve the obstacle of multiple painful daily injections at disease diagnosis, may enable pre-meal administration of insulin before meals and snacks, may improve quality of life, and most important, may decrease post prandial glucose excursions. Moreover, one should remember that children cannot decide on the amount of food prior to meal, and may need for achieving post prandial glucose in range 2 injections for each meal, one before and addition after a meal, which is hard to adhere with injections. Furthermore, toddlers receive the insulin injections after meals from fear of not finishing the meal, thus increasing significantly their post meal glycemic excursion . The early use of I-port at disease diagnosis may reduces pain, increase the amount of daily injections, may increase accuracy of insulin administration, and thus improve time in range from disease diagnosis. Previous report with Insuflon (Unomedical) showed an improvement of 0.7% in HbA1c , as well as a low rate of pain, a local response, and no blockage15, but its use is not common in the daily life of the patients in light of lack of comfort in insertion, and permission to use only one insulin type. The I-port is easier to insert and can be used in several types of insulin. The device is effective in adult population, approximately 70% to reduce the pain, about 70% improving quality of life and 70% of patients not felt in its presence, no change in HbA1c16. Its main side effect is 4% of the reported cases of local reactions16.There are no reports in the literature of the use of I-port in the pediatric population.

Technology in T1D has actually provided a solution for those multiple daily injections, by using an insulin pump 17. However, insulin pump cannot be used immediately, and not by all patients, and is not funded in many countries. Even in developed countries,asIsrael, it takes a minimum of 3 months for a patient to start using a pump in real life due to health care approvals, financial considerations, technology introduction to families, and education for the life with T1D. However, early control of glucose levels and prevention of hyperglycemic excursions was proven to prevent short and long term complications, and may lead to better long-run glycemic control .

The hypothesis is that early introduction of an I-port system, as permanent means for insulin administration, or as a bridge for future pump management, may be a simple solution in real life for multiple injections, maintaining glucose in target range and prevention of post-prandial glycemic excursions.

Aims of study:

To assess the efficacy of I-port use in recent onset T1D in a pediatric population, in increasing insulin administration and possibly improving time in range of glucose.

To compare the number of daily insulin injections, total daily insulin dose per kg, glycemic parameters, safety of administration and quality of life between multiple subcutaneous insulin injections with and without iPORT in children and adolescents with recent -onset type 1 diabetes .

Research template:

A multi-center, open label, randomized controlled clinical trial. Patients will be recruited during the first 4 weeks of diagnosis, for a study duration of 2 months.

Computerized randomization of patients will be performed to allocate them to the I-port and control groups, at a 2:1 ratio.

Use of I-port will be demonstrated and inserted for the first time to the I-port group by a diabetes nurse according to manufacture guidelines Patients will be instructed to administer insulin prior to each meal or snack according to carbohydrate counting or sliding scale.

Patients will be instructed to always use an insulin cap attached to their insulin pen Patients will use Libre continuous glucose monitoring system, as per clinical 2019 guidelines, for glucose monitoring Questionnaires regarding quality of life, treatment satisfaction and degree of pain and discomfort will be filled at end of study All participants allocated to the control group will have the opportunity to use I-port for 2 months at end of study, with no cost.

All study equipment, including insulin caps and activity tracker will remain at participants possession at end of study.

Research duration:

The study is anticipated to last approximately 24 months from first investigational center initiation to finalization of all data entry and monitoring procedures. Subject participation is expected to be approximately of 60 days.

Study population:

The study population will include 35 patients (according to sample size calculation, as described below) aged 1-18 years with type 1 diabetes

Non-investigational Additional Devices:

1. Abbott Libre Flash Glucose Monitoring https://www.diabetescare.abbott/worldwide-locations.html
2. Dexcom CGM sensor system https://www.dexcom.com/get-started-cgm/ Both systems are continuous glucose monitoring systems, used for clinical care according to guidelines and ministry of health approved devices for T1D management since January 2020 or all T1DM patients
3. Smart Insulin Pen Cap - Clipsulin™* (Diabnext) to capture by bluetooth connecter all administered insulin doses including their time and dose, and food if logged in. This is the only current novel mean available to capture real time accurate insulin administration by patients. All data will be collected by an app. We will use in this study a device DiabNext Clipsulin: https://www.diabnext.com/clipsulin-c3/

2. Fitbit™* Fitness Tracker or Apple Watch™* HealthKit™. An activity tracker, which will be used in order to catch movement according to food, and insulin administration. This is not a medical device, looks like a watch.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes within the last 4 weeks
* Need for insulin injections at least 1 times a day
* Age of 1-18 years.
* Agree to comply with all the terms of the study
* Has an iPhone, iOS 11 or higher OR Android

Exclusion Criteria:

* Insulin pump therapy

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Daily insulin administration per day | 2 years
  The difference in number of insulin administrations per day between I-port and control groups
Total insulin daily dose per kg per day | 2 years
  The difference in total daily insulin dose per kg per day between I-port and control groups

SECONDARY OUTCOMES:
Time in Range difference | 2 years
  The difference in time in range of glucose per day between I-port and control groups
hyperglycemic and hypoglycemic ranges of glucose per day | 2 years
  The difference in time in hyperglycemic and hypoglycemic ranges of glucose per day between I-port and control groups
HbA1c | 2 years
  The change in HbA1c from baseline to end of study between I-port and control groups
coefficient of variability (CV) | 2 years
  The difference in coefficient of variability (CV) between I-port and control groups
quality of life difference scale 1-46, higher is better | 2 years
  quality of life difference as measured by PedsQL questionnaire
treatment satisfaction, scale up to 10, higher is better | 2 years
  treatment satisfaction as measured by DTSQ questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Avital Leshem, Study Director — Assaf-Harofeh Medical Center

IPD SHARING:
Plan to Share IPD: No